CLINICAL TRIAL: NCT06879964
Title: Usefulness of Post-Operative Radiotherapy in High-grade Cutaneous Squamous Cell Carcinoma: an Observational Study
Acronym: PORTSCC
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Chiara Giorgini, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: PORTSCC
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Cutaneous Squamous Cell Carcinoma (CSCC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with high-grade cutaneous squamous cell carcinoma

SUMMARY:
Post-operative radiotherapy (PORT) is currently considered as the second most important therapy to treat high-grade cutaneous squamous cell carcinoma. Nonetheless, only few studies evaluate its impact on recurrence rate and the major part of those ones do not include a proper control group of patients.

Most recent guide lines from NCCN, Sidemast and British associations of dermatologists suggest clinicians to offer or consider PORT in selected patients but class nor level of evidence of those guide lines are provided.

This project evaluates impact of post-operative radiotherapy on recurrence rate and overall survival by comparing two cohort of patients, the former who accepted PORT and the latter who, nonetheless its necessity, decided to not undergo it.

The hypothesis which this project will answer concerns the effectiveness of post-operative radiotherapy in preventing local and regional recurrences. We expect a significant decrease of recurrence rate in patients who undergo this therapeutic option as compared to those with clinical indication but do not undergo PORT.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of high-grade cutaneous squamous cell carcinoma
* patients eligible for post-operative radiotherapy
* minimum follow-up of 24 months

Exclusion Criteria:

* lack of clinical of histological data
* impossibility of a proper follow-up
* occurrence of intermediate events (i.e., pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of high-grade cutaneous squamous cell carcinoma, eligible for post-operative radiotherapy, cared for at the Dermatologic Clinic, Fondazione IRCCS Policlinico San Matteo.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
effectiveness of post-operative radiotherapy in preventing local and regional recurrences | 24 months
  Association of PORT and recurrence rate, considering PORT as a binary variable (yes/no) and evaluating recurrence with a clinical and echographic follow-up with a minimum duration of 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Dermatologia, Pavia, Pavia, Italy